CLINICAL TRIAL: NCT07317245
Title: HUmanitas PROtontherapy (HU-PRO)
Acronym: HU-PRO
Status: Recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: PRO/OSS - 001/2026
Record Dates: First submitted 2025-12-18; First posted 2026-01-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Proton Therapy
Keywords: registry; cancer; proton therapy; re-irradiation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- proton therapy: all patients treated with proton therapy according to clinical practice

SUMMARY:
Proton therapy is a cancer treatment, similar to the more commonly used radiation therapy. It uses radiation to destroy cancer cells and helps control the disease in the treated area.

However, when proton therapy is compared with standard radiation therapy, many studies show fewer side effects and better disease control. This is due to the unique physical properties of the particles used in proton therapy.

At present, in Italy, this innovative treatment is available only for selected diseases, as defined by national guidelines. For this reason, it is very important to collect as much data as possible to support the further development of proton therapy and to improve treatment safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumors candidate to proton therapy, in particular, according to Italian regolamentations
* Written informed consent for HU-PRO according to applicable legal and ethical requirements
* Indication for proton therapy
* ≥ 18 years old
* ECOG PS (performance status scale) 0-2

Exclusion Criteria:

* Age < 18 years old
* ECOG (performance status scale) >3
* Life expectancy < 3 months
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with indication to proton therapy treatment
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2036-01 (Estimated); Study Completion 2036-01 (Estimated)

PRIMARY OUTCOMES:
collecting real world data | from enrollment to 10 years
  To collect real-world data on cancer patients treated with protonherapy, to support research and to provide evidence of the role of protontherapy in a multidisciplinary approach.

SECONDARY OUTCOMES:
toxicities profiles | from enrollment to 10 years
  Asses acute and late onset side effects and compare toxicity rates with conventional radiotherapy (toxicity classification by CTCAE)
identify prognostic biomarkers | from enrollment to 10 years
  Investigate biological and clinical factors that influence treatment response and survival (blood samples and saliva samples for Head&Neck patients)
Optimize treatment plannig | from enrollment to 10 years
  Asses different proton therapy techniques and procedures to refine clinical practice (Radiotherapy plans comparison)
Secondary Cancer Risk | from enrollment to 10 years
  Monitoring long term cancer incidence in patients treated with proton therapy, especially in young patients (clinical data comparison - appearance of disease after treatment)
Asses Outcomes in Rare or Radioresistant Tumors | from enrollment to 10 years
  Collect data on tumor types with limited evidence to determine optimal indications for proton therapy (clinical data comparison)
Monitor Treatment Adherence and Compliance | from enrollment to 10 years
  Evaluate factors influencing patient adherence to treatment schedules and follow up care
Analyze Quality of Life Outcomes | from enrollment to 10 years
  Measure patient reported outcomes (PROs) to understand the impact of proton therapy on daily life and well being (QLQ-C30 and different questionnaries according to pathology site)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Humanitas Research Hospital, Rozzano, Michigan, Italy